CLINICAL TRIAL: NCT03239522
Title: An Open-label Study in Healthy Male Participants to Determine the Mass Balance, Absolute Bioavailability and Pharmacokinetics of Daprodustat, Administered as a Single Intravenous Microtracer (Concomitant With an Oral Dose of Non-radiolabelled Daprodustat) and a Single, Oral Radiolabelled Dose
Brief Title: Absorption and Elimination of Radiolabeled Daprodustat
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 200232; 2017-001729-42 (EudraCT Number)
Record Dates: First submitted 2017-07-17; First posted 2017-08-04 (Actual); Results first posted 2019-03-18 (Actual); Last update posted 2019-12-03 (Actual); Status verified 2019-11

CONDITIONS: Anaemia
Keywords: GSK1278863; pharmacokinetics; mass balance; daprodustat
MeSH Terms: conditions — Anemia | interventions — Infusions, Intravenous; GSK1278863; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- All participants receiving treatment (Experimental): Each participant will receive a single 6 milligram (mg) oral dose of daprodustat on Day 1 of period 1. After approximately 1 hour, participants will receive 50 microgram (µg) of [14C]-GSK1278863 by IV infusion over 1 hour. On Day 1 of period 2, each participant will receive 25 mg [14C]-GSK1278863 as an oral solution.
  Interventions: Drug: [14C]-GSK1278863 solution for IV infusion; Drug: [14C]-GSK1278863 oral solution; Drug: Daprodustat 6 mg oral tablet

INTERVENTIONS:
Drug: [14C]-GSK1278863 solution for IV infusion — It is a clear, colorless solution free from visible particulate matter. Participants will receive 10 mL of 5 µg/mL of [14C]-GSK1278863 IV solution (total dose: 50 µg) by IV infusion over 1 hour.
Drug: [14C]-GSK1278863 oral solution — It is a clear, colorless solution. Participants will receive 125 mL of 200 µg/mL of [14C]-GSK1278863 oral solution (total dose: 25 mg).
Drug: Daprodustat 6 mg oral tablet — It is a 9.0 millimeter (mm) round, white film coated tablet.

SUMMARY:
Absorption, metabolism and excretion of daprodustat (GSK1278863) have been studied in previous clinical trials; however, the elimination routes and metabolic pathways of daprodustat have not been fully elucidated in humans. This is an open-label, single-center, non-randomized, 2-period, single-sequence, crossover, mass balance study in 6 healthy male participants. The aim of the study is to assess the excretion balance of daprodustat using [14C]-radiolabeled drug substance administered orally, and as an intravenous (IV) infusion, administered as a microtracer dose (concomitant with an oral, non-radiolabeled dose). Absolute bioavailability of an oral dose will also be assessed. Each participant will be involved in the study for up to 10 weeks which include a screening visit, two treatment periods (treatment periods 1 and 2), separated by about 7 days (at least 14 days between oral doses), and a follow up visit 1-2 weeks after the last assessment in treatment period 2. The primary objective of the study is to gain a better understanding of the compound's excretory and metabolic profile. This study will include sampling of duodenal bile to conduct qualitative assessment of drug metabolites in this matrix in order to characterize biliary elimination pathways.

ELIGIBILITY:
Inclusion Criteria:

* Aged 30 to 55 years, inclusive, at the time of signing the informed consent.
* Healthy, as determined by the investigator or medically qualified designee, based on a medical evaluation including medical history, physical examination, vital signs, laboratory tests, and ECG. A participant with a clinical abnormality or laboratory parameter (i.e., outside the reference range for the population being studied), which is not specifically listed in the eligibility criteria, may be included only if the investigator agrees and documents that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Hemoglobin value at screening greater than the lower limit of the laboratory reference range and less than or equal to 16.0 gram (g) per deciliter (dL).
* History of regular bowel movements (averaging one or more bowel movements per day).
* Non-smoker, or ex-smoker who hasn't regularly smoked for the 6 months before screening.
* Body weight of 50 kilogram (kg) and above, and body mass index (BMI) within the range 19.0-31 kg per meter (m)^2 (inclusive).
* Participants must agree to use contraception as follows: participants with female partners of childbearing potential must agree to use a condom from the time of first dose of study treatment until 1 month after their last dose.
* Capable of giving signed informed consent.
* Willingness to give written consent to have data entered into The Over-volunteering Prevention System.

Exclusion Criteria:

* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones). Participants with a history of cholecystectomy must be excluded.
* Any clinically relevant abnormality identified at the screening medical assessment (physical examination/medical history), clinical laboratory tests, or 12-lead ECG.
* Myocardial infarction or acute coronary syndrome <=12 weeks prior to screening through to enrollment (Day 1, treatment period 1).
* History or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal (GI), endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs, or which could constitute a risk when taking the study treatment, or interfere with the interpretation of data.
* Evidence of actively bleeding gastric, duodenal or esophageal ulcer disease OR clinically significant GI bleeding <=12 weeks prior to screening through to enrollment (Day 1, treatment period 1).
* History of malignancy within the two years before dosing, with the exception of localized squamous cell or basal cell carcinoma of the skin that has been definitively treated prior to screening; currently receiving treatment for cancer; has a strong family history of cancer (e.g., familial cancer disorders).
* Mentally or legally incapacitated.
* Heart Failure: Class II, III or IV heart failure, as defined by the New York Heart Association (NYHA) functional classification system.
* Any other condition, clinical or laboratory abnormality, or examination finding that the investigator considers would put the participant at unacceptable risk, which may affect study compliance or prevent understanding of the aims or investigational procedures or possible consequences of the study.
* Daprodustat is a substrate of cytochrome P4502C8 (CYP2C8). Co-administration of drugs that are inhibitors of this enzyme are prohibited.
* Past or intended use of over-the-counter or prescription medication including herbal medications prior to dosing except occasional use of paracetamol (acetaminophen), within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study treatment until completion of the follow-up visit, unless in the opinion of the investigator and GSK medical monitor the medication will not interfere with the study.
* Current enrolment in a clinical trial; recent participation in a clinical trial and has received an investigational product within 3 months before their first dose in the current study.
* Exposure to more than 4 new chemical entities within 12 months before their first dose in the current study.
* Participation in a clinical trial involving administration of 14C-labelled compound(s) within the last 12 months. A participant's previous effective dose will be reviewed by the medical investigator to ensure there is no risk of contamination/carryover into the current study.
* Received a total body radiation dose of greater than 10.0 millisievert (mSv) (upper limit of world health organization [WHO] category II) or exposure to significant radiation (e.g., serial x-ray or computed tomography [CT] scans, barium meal, etc.) in the 3 years before this study.
* Alanine transaminase (ALT) >1.5 times upper limit of normal (ULN).
* Bilirubin >1.5 times ULN (isolated bilirubin >1.5 times ULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* QTc >500 millisecond (msec). The QTc must be the QTcB.
* Presence of Hepatitis B surface antigen (HBsAg) at screening or positive Hepatitis C antibody test result at screening or within 3 months before the first dose of study treatment.
* Positive pre-study drug/alcohol screen.
* Positive human immunodeficiency virus (HIV) antibody test.
* Regular use of known drugs of abuse.
* Regular alcohol consumption within 6 months prior to the study defined as an average weekly intake of >21 units. One unit is equivalent to 8 g of alcohol: a glass (approximately 240 milliliter [mL]) of beer, 1 small glass (approximately 100 mL) of wine or 1 (approximately 25 mL) measure of spirits.
* At screening, a supine blood pressure (BP) that is persistently higher than 140/90 millimeters of mercury (mmHg) taken in triplicate, unless deemed not clinically significant by the investigator.
* At screening, a supine mean heart rate (HR) outside the range of 40-100 beats per minute, unless deemed not clinically significant by the investigator.
* Has had an occupation which requires monitoring for radiation exposure, nuclear medicine procedures, or excessive x-rays within the past 12 months.
* Unable to refrain from consumption of prohibited food and drinks from 7 days before the first dose of study medication until the follow up visit.
* Participation in the study would result in donation of blood or blood products in excess of 550 mL within a 90 day period.
* Unwillingness or inability to follow the procedures, including the use of the Entero-Test capsule.
* Urinary cotinine levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products in the 6 months prior to screening.
* History of drug abuse or dependence within 6 months of the study.
* History of sensitivity to daprodustat, or their components thereof, or a history of drug or other allergy that, in the opinion of the investigator or GSK medical monitor, contraindicates their participation.

Ages: 30 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only male participants, aged 30 to 55 years (inclusive) will be enrolled into the study.
Enrollment: 6 (Actual)
Dates: Start 2017-10-10 (Actual); Primary Completion 2017-11-28 (Actual); Study Completion 2017-11-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study evaluated the excretion balance of daprodustat(GSK1278863) using radiolabeled 14 Carbon [14C]-drug substance administered orally, and as an intravenous (IV) infusion, administered as a micro tracer dose (concomitant with an oral, non-radiolabeled dose) in healthy male participants.
Pre-assignment Details: Participants were enrolled at a single center in United Kingdom. A total of 6 participants were enrolled in the study. All the enrolled participants were randomized to receive study treatment.
Groups:
- All Participants Receiving GSK1278863: Participants received a single 6 milligram (mg) oral dose of GSK1278863 on Day 1 of treatment period 1, after an overnight fast of at least 8 hours. After approximately 1 hour, participants received 50 microgram (µg) [14C]-GSK1278863 by IV infusion over 1 hour. It was followed by a washout period of 7 days. On Day 1 of treatment period 2, each participant received 25 mg [14C]-GSK1278863 as an oral solution, after an overnight fast of at least 8 hours.
Period: Treatment Period 1 (Up to 7 Days)
Arm/Group | All Participants Receiving GSK1278863
Started | 6
Completed | 6
Not Completed | 0
Period: Washout Period (Up to 7 Days)
Arm/Group | All Participants Receiving GSK1278863
Started | 6
Completed | 6
Not Completed | 0
Period: Treatment Period 2 (Up to 15 Days)
Arm/Group | All Participants Receiving GSK1278863
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Participants Receiving GSK1278863
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: Years] | 40.7 (8.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  WHITE - ARABIC/NORTH AFRICAN HERITAGE | 1
  WHITE - WHITE/CAUCASIAN/EUROPEAN HERITAGE | 5

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve From Time Zero (Pre-dose) Extrapolated to Infinite Time (AUC [0-Inf]) of Total Drug-related Material (Radioactivity) in Plasma Following Administration of GSK1278863
Description: Plasma samples were collected from participants at indicated time points in each of the treatment period 1 and 2, after administration of study treatment to investigate the pharmacokinetics of GSK1278863 in plasma. Pharmacokinetic analysis was conducted using standard non-compartmental methods. Pharmacokinetic Population comprised of all participants in the Safety Population who had at least 1 non-missing pharmacokinetic assessment (Non-quantifiable [NQ] values were considered as non-missing values).
Time Frame: Pre-dose, 0.5, 1, 1.25, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120 and 144 hours post-dose in treatment period 1; Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120 and 144 hours post-dose in treatment period 2
Population: Pharmacokinetic Population. Only those participants with data available at specified time point were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*nanogram equivalent per milliliter
Groups:
- [14C]-GSK1278863 50 µg IV Infusion: Participants received 50 µg [14C]-GSK1278863 by IV infusion over 1 hour in treatment period 1, after approximately 1 hour of receiving GSK1278863 6 mg Oral tablet.
- [14C]-GSK1278863 25 mg Oral Solution: Participants received 25 mg [14C]-GSK1278863 as an oral solution, after an overnight fast of at least 8 hours in treatment period 2.
Arm/Group | [14C]-GSK1278863 50 µg IV Infusion | [14C]-GSK1278863 25 mg Oral Solution
Number analyzed (Participants) | 5 | 6
Hour*nanogram equivalent per milliliter | 6.6864 (19.8) | 2278.8914 (18.2)

2. Primary Outcome: AUC (0-Inf) of Total Drug-related Material (Radioactivity) in Blood Following Administration of GSK1278863
Description: Blood samples were planned to be collected from participants at indicated time points in each of the treatment period 1 and 2, after administration of study treatment to investigate the pharmacokinetics of GSK1278863 in blood. Data were not collected for blood total radioactivity concentration following administration of radiolabeled IV dose of GSK1278863 because of an error (deviation). The deviation is due to a processing error: labels for whole blood draws, and aliquots for shipment were not generated in error. Data were not analyzed for radiolabeled oral dose of GSK1278863 as there were not enough data points captured for a terminal slope required to calculate AUC (0-inf). The blood assay could not detect radiation levels at the time points blood was drawn to go into these calculations.
Time Frame: as for outcome 1
Population: Pharmacokinetic Population. Data were not collected for radiolabeled IV dose of GSK1278863 because of an error (deviation). Data were not analyzed for radiolabeled oral dose GSK1278863 as there were not enough data points captured for a terminal slope required to calculate AUC (0-inf).
Arm/Group | [14C]-GSK1278863 50 µg IV Infusion | [14C]-GSK1278863 25 mg Oral Solution
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: AUC From Time Zero (Pre-dose) to Last Time of Quantifiable Concentration Within a Participant Across All Treatments (AUC [0-t]) of Total Drug-related Material (Radioactivity) in Plasma Following Administration of GSK1278863
Description: Plasma samples were collected from participants at indicated time points in each of the treatment period 1 and 2, after administration of study treatment to investigate the pharmacokinetics of GSK1278863 in plasma. Pharmacokinetic analysis was conducted using standard non-compartmental methods.
Time Frame: as for outcome 1
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*nanogram equivalent per milliliter
Arm/Group | [14C]-GSK1278863 50 µg IV Infusion | [14C]-GSK1278863 25 mg Oral Solution
Number analyzed (Participants) | 6 | 6
Hour*nanogram equivalent per milliliter | 6.5252 (18.9) | 2206.7099 (18.5)

4. Primary Outcome: AUC (0-t) of Total Drug-related Material (Radioactivity) in Blood Following Administration of GSK1278863
Description: Blood samples were collected from participants at indicated time points after administration of study treatment to investigate the pharmacokinetics of GSK1278863 in blood. Pharmacokinetic analysis was conducted using standard non-compartmental methods. Data were not collected for blood total radioactivity concentration following administration of radiolabeled IV dose of GSK1278863 because of an error (deviation). The deviation is due to a processing error: labels for whole blood draws, and aliquots for shipment were not generated in error.
Time Frame: as for outcome 1
Population: Pharmacokinetic Population. Data were not collected for radiolabeled IV dose of GSK1278863 because of an error (deviation).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*nanogram equivalent per milliliter
Arm/Group | [14C]-GSK1278863 50 µg IV Infusion | [14C]-GSK1278863 25 mg Oral Solution
Number analyzed (Participants) | 0 | 6
Hour*nanogram equivalent per milliliter |  | 824.6102 (17.2)

5. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Total Drug-related Material (Radioactivity) in Plasma Following Administration of GSK1278863
Description: as for outcome 3
Time Frame: as for outcome 1
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram equivalent per milliliter
Arm/Group | [14C]-GSK1278863 50 µg IV Infusion | [14C]-GSK1278863 25 mg Oral Solution
Number analyzed (Participants) | 6 | 6
Nanogram equivalent per milliliter | 3.0114 (15.8) | 623.9059 (34.8)

6. Primary Outcome: Cmax of Total Drug-related Material (Radioactivity) in Blood Following Administration of GSK1278863
Description: as for outcome 4
Time Frame: as for outcome 1
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram equivalent per milliliter
Arm/Group | [14C]-GSK1278863 50 µg IV Infusion | [14C]-GSK1278863 25 mg Oral Solution
Number analyzed (Participants) | 0 | 6
Nanogram equivalent per milliliter |  | 289.9998 (30.7)

7. Primary Outcome: Time of Occurrence of Cmax (Tmax) of Total Drug-related Material (Radioactivity) in Plasma Following Administration of GSK1278863
Description: as for outcome 3
Time Frame: as for outcome 1
Population: Pharmacokinetic Population
Measure: Median (Full Range); unit: Hour
Arm/Group | [14C]-GSK1278863 50 µg IV Infusion | [14C]-GSK1278863 25 mg Oral Solution
Number analyzed (Participants) | 6 | 6
Hour | 0.9833 [0.983 to 1.250] | 0.7583 [0.500 to 3.000]

8. Primary Outcome: Tmax of Total Drug-related Material (Radioactivity) in Blood Following Administration of GSK1278863
Description: as for outcome 4
Time Frame: as for outcome 1
Population: as for outcome 4
Measure: Median (Full Range); unit: Hour
Arm/Group | [14C]-GSK1278863 50 µg IV Infusion | [14C]-GSK1278863 25 mg Oral Solution
Number analyzed (Participants) | 0 | 6
Hour |  | 1.0000 [1.000 to 3.000]

9. Primary Outcome: Apparent Terminal Phase Half-life (t1/2) of Total Drug-related Material (Radioactivity) in Plasma Following Administration of GSK1278863
Description: as for outcome 3
Time Frame: as for outcome 1
Population: Pharmacokinetic Population. Only those participants with data available at specified time point were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour
Arm/Group | [14C]-GSK1278863 50 µg IV Infusion | [14C]-GSK1278863 25 mg Oral Solution
Number analyzed (Participants) | 5 | 6
Hour | 6.7699 (106.4) | 61.8251 (15.1)

10. Primary Outcome: T1/2 of Total Drug-related Material (Radioactivity) in Blood Following Administration of GSK1278863
Description: Blood samples were planned to be collected from participants at indicated time points in each of the treatment period 1 and 2, after administration of study treatment to investigate the pharmacokinetics of GSK1278863 in blood. Data were not collected for blood total radioactivity concentration following administration of radiolabeled IV dose of GSK1278863 because of an error (deviation). The deviation is due to a processing error: labels for whole blood draws, and aliquots for shipment were not generated in error. Data were not analyzed for radiolabeled oral dose of GSK1278863 as there were not enough data points captured for a terminal slope required to calculate t1/2. The blood assay could not detect radiation levels at the time points blood was drawn to go into these calculations.
Time Frame: as for outcome 1
Population: Pharmacokinetic Population. Data were not collected for radiolabeled IV dose of GSK1278863 because of an error (deviation). Data were not analyzed for radiolabeled oral dose GSK1278863 as there were not enough data points captured for a terminal slope required to calculate t1/2.
Arm/Group | [14C]-GSK1278863 50 µg IV Infusion | [14C]-GSK1278863 25 mg Oral Solution
Number analyzed (Participants) | 0 | 0

11. Primary Outcome: Volume of Distribution at Steady State (Vss) of Total Drug-related Material (Radioactivity) in Plasma Following IV Dose of GSK1278863
Description: Plasma samples were collected from participants at indicated time points in treatment period 1, after administration of study treatment to investigate the pharmacokinetics of GSK1278863 in plasma. Pharmacokinetic analysis was conducted using standard non-compartmental methods.
Time Frame: Pre-dose, 0.5, 1, 1.25, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120 and 144 hours post-dose in treatment period 1
Population: Pharmacokinetic Population. Only those participants with data available at specified time point were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | [14C]-GSK1278863 50 µg IV Infusion
Number analyzed (Participants) | 5
Liters | 32.2355 (59.1)

12. Primary Outcome: Vss of Total Drug-related Material (Radioactivity) in Blood Following IV Dose of GSK1278863
Description: Blood samples were planned to be collected from participants at indicated time points in treatment period 1, after administration of study treatment to investigate the pharmacokinetics of GSK1278863 in blood. Data were not collected for blood total radioactivity concentration following administration of radiolabeled IV dose of GSK1278863 because of an error (deviation). The deviation is due to a processing error: labels for whole blood draws, and aliquots for shipment were not generated in error.
Time Frame: as for outcome 11
Population: as for outcome 4
Arm/Group | [14C]-GSK1278863 50 µg IV Infusion
Number analyzed (Participants) | 0

13. Primary Outcome: Total Systemic Clearance (CL) of Total Drug-related Material (Radioactivity) in Plasma Following IV Dose of GSK1278863
Description: Plasma samples were collected from participants at indicated time points in treatment period 1 after administration of study treatment to investigate the pharmacokinetics of GSK1278863 in plasma. Pharmacokinetic analysis was conducted using standard non-compartmental methods.
Time Frame: as for outcome 11
Population: Pharmacokinetic Population. Only those participants with data available at specified time point were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters per hour
Arm/Group | [14C]-GSK1278863 50 µg IV Infusion
Number analyzed (Participants) | 5
Liters per hour | 7.4779 (19.8)

14. Primary Outcome: CL of Total Drug-related Material (Radioactivity) in Blood Following IV Dose of GSK1278863
Description: Blood samples were planned to be collected from participants at indicated time points in treatment period 1 after administration of study treatment to investigate the pharmacokinetics of GSK1278863 in blood. Data were not collected for blood total radioactivity concentration following administration of radiolabeled IV dose of GSK1278863 because of an error (deviation). The deviation is due to a processing error: labels for whole blood draws, and aliquots for shipment were not generated in error.
Time Frame: as for outcome 11
Population: as for outcome 4
Arm/Group | [14C]-GSK1278863 50 µg IV Infusion
Number analyzed (Participants) | 0

15. Primary Outcome: Percentage of the Total Radioactive Dose Excreted in Urine Over Time Following a Single, Oral Dose of [14C]-GSK1278863
Description: Urine samples were collected at the indicated time points to determine the rate and extent of excretion of total radioactivity in urine. All participants were asked to void their bladders before study treatment administration.
Time Frame: Pre-dose and then over 24 hours collection periods as follows: 0-24, 24-48, 48-72, 72-96, 96-120,120-144 and 144-168 hours post-dose in treatment period 2
Population: Pharmacokinetic Population. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Measure: Mean (Standard Deviation); unit: Percent dose excreted
Arm/Group | [14C]-GSK1278863 25 mg Oral Solution
Number analyzed (Participants) | 6
Percent dose excreted
  Pre-dose; n=6 | 0.000 (0.0000)
  0-24 hours; n=6 | 20.450 (2.7441)
  24-48 hours; n=6 | 20.838 (2.8280)
  48-72 hours; n=6 | 21.003 (2.8723)
  72-96 hours; n=6 | 21.065 (2.8744)
  96-120 hours; n=6 | 21.065 (2.8744)
  120-144 hours; n=6 | 21.065 (2.8744)
  144-168 hours; n=5: number analyzed (Participants) | 5
  144-168 hours; n=5 | 21.434 (3.0507)

16. Primary Outcome: Percentage of the Total Radioactive Dose Excreted in Feces Over Time Following a Single, Oral Dose of [14C]-GSK1278863
Description: Fecal samples were collected at the indicated time points to determine the rate and extent of excretion of total radioactivity in feces.
Time Frame: Pre-dose and then over 24 hour collection periods as follows: 0-24, 24-48, 48-72, 72-96, 96-120, 120-144 and 144-168 hours post-dose in treatment period 2
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: Percent dose excreted
Arm/Group | [14C]-GSK1278863 25 mg Oral Solution
Number analyzed (Participants) | 6
Percent dose excreted
  Pre-dose; n=6 | 0.000 (0.0000)
  0-24 hours; n=5: number analyzed (Participants) | 5
  0-24 hours; n=5 | 0.096 (0.1292)
  24-48 hours; n=5: number analyzed (Participants) | 5
  24-48 hours; n=5 | 22.298 (31.0164)
  48-72 hours; n=6 | 49.988 (25.3857)
  72-96 hours; n=6 | 68.312 (6.0872)
  96-120 hours; n=5: number analyzed (Participants) | 5
  96-120 hours; n=5 | 73.450 (3.1046)
  120-144 hours; n=5: number analyzed (Participants) | 5
  120-144 hours; n=5 | 74.698 (2.1027)
  144-168 hours; n=4: number analyzed (Participants) | 4
  144-168 hours; n=4 | 73.553 (3.6611)

17. Primary Outcome: Percentage of the Total Radioactive Dose Excreted in Urine and Feces Determined as Total Excretion Over Time
Description: Urine and fecal samples were collected at the indicated time points to determine the rate and extent of cumulative excretion of total radioactivity in urine and feces.
Time Frame: as for outcome 16
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: Percent dose excreted
Arm/Group | [14C]-GSK1278863 25 mg Oral Solution
Number analyzed (Participants) | 6
Percent dose excreted
  Pre-dose; n=6 | 0.000 (0.0000)
  0-24 hours; n=6 | 20.530 (2.7223)
  24-48 hours; n=6 | 39.433 (28.2968)
  48-72 hours; n=6 | 70.992 (25.9980)
  72-96 hours; n=6 | 89.377 (6.3351)
  96-120 hours; n=6 | 94.177 (2.1428)
  120-144 hours; n=6 | 94.705 (2.0982)
  144-168 hours; n=5: number analyzed (Participants) | 5
  144-168 hours; n=5 | 94.582 (2.3066)

18. Secondary Outcome: AUC (0-Inf) of GSK1278863 in Plasma Following Administration IV and Both Oral Doses
Description: Plasma samples were collected from participants at indicated time points, after administration of IV dose, both radiolabeled and non-radiolabeled oral doses of GSK1278863. Pharmacokinetic analysis was conducted using standard non-compartmental methods.
Time Frame: as for outcome 1
Population: Pharmacokinetic Population. Only those participants with data available at specified time point were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*nanogram per milliliter
Groups:
- GSK1278863 6 mg Oral Tablet: Participants received a single 6 mg oral tablet of GSK1278863 on Day 1 of treatment period 1, after an overnight fast of at least 8 hours.
Arm/Group | GSK1278863 6 mg Oral Tablet | [14C]-GSK1278863 50 µg IV Infusion | [14C]-GSK1278863 25 mg Oral Solution
Number analyzed (Participants) | 6 | 3 | 6
Hour*nanogram per milliliter | 199.2552 (16.9) | 2.6509 (27.4) | 940.2011 (28.6)

19. Secondary Outcome: AUC(0-t) of GSK1278863 in Plasma Following Administration of IV and Both Oral Doses
Description: as for outcome 18
Time Frame: as for outcome 1
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*nanogram per milliliter
Arm/Group | GSK1278863 6 mg Oral Tablet | [14C]-GSK1278863 50 µg IV Infusion | [14C]-GSK1278863 25 mg Oral Solution
Number analyzed (Participants) | 6 | 6 | 6
Hour*nanogram per milliliter | 198.1658 (16.8) | 2.6368 (20.4) | 938.5541 (28.7)

20. Secondary Outcome: Cmax of GSK1278863 in Plasma Following Administration of IV and Both Oral Doses
Description: as for outcome 18
Time Frame: as for outcome 1
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | GSK1278863 6 mg Oral Tablet | [14C]-GSK1278863 50 µg IV Infusion | [14C]-GSK1278863 25 mg Oral Solution
Number analyzed (Participants) | 6 | 6 | 6
Nanogram per milliliter | 96.1190 (17.2) | 2.0058 (25.5) | 544.7022 (34.1)

21. Secondary Outcome: Tmax of GSK1278863 in Plasma Following Administration of IV and Both Oral Doses
Description: as for outcome 18
Time Frame: as for outcome 1
Population: Pharmacokinetic Population
Measure: Median (Full Range); unit: Hour
Arm/Group | GSK1278863 6 mg Oral Tablet | [14C]-GSK1278863 50 µg IV Infusion | [14C]-GSK1278863 25 mg Oral Solution
Number analyzed (Participants) | 6 | 6 | 6
Hour | 2.1167 [1.417 to 4.000] | 0.983 [0.983 to 0.983] | 0.5000 [0.500 to 0.517]

22. Secondary Outcome: T1/2 of GSK1278863 in Plasma Following Administration of IV and Both Oral Doses
Description: as for outcome 18
Time Frame: as for outcome 1
Population: Pharmacokinetic Population. Only those participants with data available at specified time point were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour
Arm/Group | GSK1278863 6 mg Oral Tablet | [14C]-GSK1278863 50 µg IV Infusion | [14C]-GSK1278863 25 mg Oral Solution
Number analyzed (Participants) | 6 | 3 | 6
Hour | 1.8786 (21.6) | 2.0653 (6.6) | 2.5037 (30.2)

23. Secondary Outcome: AUC (0-Inf) of GSK1278863 Metabolites in Plasma Following Administration of IV and Both Oral Doses
Description: Plasma samples were collected from participants at indicated time points, for metabolite profiling. GSK2391220, GSK2506104, GSK2487818, GSK2506102, GSK2531398 and GSK2531401 were metabolites of GSK1278863.Pharmacokinetic analysis was conducted using standard non-compartmental methods. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles). Data were not collected for GSK1278863 metabolites following IV dose as analysis of pharmacokinetic parameters of only parent compound following IV dose was of interest to calculate the bioavailability and not the metabolites.
Time Frame: as for outcome 1
Population: Pharmacokinetic Population. Data were not collected for GSK1278863 metabolites following IV dose as analysis of pharmacokinetic parameters of only parent compound following IV dose was of interest to calculate the bioavailability and not the metabolites.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*nanogram per milliliter
Arm/Group | GSK1278863 6 mg Oral Tablet | [14C]-GSK1278863 50 µg IV Infusion | [14C]-GSK1278863 25 mg Oral Solution
Number analyzed (Participants) | 6 | 0 | 6
Hour*nanogram per milliliter
  GSK2391220; n=6,0,5: number analyzed (Participants) | 6 | 0 | 5
  GSK2391220; n=6,0,5 | 33.7699 (15.1) |  | 139.7713 (19.0)
  GSK2487818; n=6,0,6 | 21.7209 (16.3) |  | 92.0554 (16.7)
  GSK2506102; n=6,0,6 | 8.6207 (15.5) |  | 33.1332 (15.6)
  GSK2506104; n=6,0,5: number analyzed (Participants) | 6 | 0 | 5
  GSK2506104; n=6,0,5 | 34.1180 (11.9) |  | 140.3785 (16.7)
  GSK2531398; n=6,0,6 | 15.0285 (13.1) |  | 61.7760 (15.4)
  GSK2531401; n=6,0,6 | 34.4699 (21.9) |  | 124.1320 (25.5)

24. Secondary Outcome: AUC(0-t) of GSK1278863 Metabolites in Plasma Following Administration of IV and Both Oral Doses
Description: Plasma samples were collected from participants at indicated time points, for metabolite profiling. GSK2391220, GSK2506104, GSK2487818, GSK2506102, GSK2531398 and GSK2531401 were metabolites of GSK1278863. Pharmacokinetic analysis was conducted using standard non-compartmental methods. Data were not collected for GSK1278863 metabolites following IV dose as analysis of pharmacokinetic parameters of only parent compound following IV dose was of interest to calculate the bioavailability and not the metabolites.
Time Frame: as for outcome 1
Population: as for outcome 23
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*nanogram per milliliter
Arm/Group | GSK1278863 6 mg Oral Tablet | [14C]-GSK1278863 50 µg IV Infusion | [14C]-GSK1278863 25 mg Oral Solution
Number analyzed (Participants) | 6 | 0 | 6
Hour*nanogram per milliliter
  GSK2391220 | 32.2574 (15.0) |  | 142.2907 (18.9)
  GSK2487818 | 21.2933 (16.8) |  | 90.9953 (16.7)
  GSK2506102 | 8.0798 (14.1) |  | 31.8897 (15.9)
  GSK2506104 | 32.3120 (11.9) |  | 142.3372 (15.6)
  GSK2531398 | 14.4743 (13.4) |  | 60.2615 (15.5)
  GSK2531401 | 31.7836 (18.8) |  | 122.7102 (25.8)

25. Secondary Outcome: Cmax of GSK1278863 Metabolites in Plasma Following Administration of IV and Both Oral Doses
Description: as for outcome 24
Time Frame: as for outcome 1
Population: Pharmacokinetic Population.Data were not collected for GSK1278863 metabolites following IV dose as analysis of pharmacokinetic parameters of only parent compound following IV dose was of interest to calculate the bioavailability and not the metabolites.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | GSK1278863 6 mg Oral Tablet | [14C]-GSK1278863 50 µg IV Infusion | [14C]-GSK1278863 25 mg Oral Solution
Number analyzed (Participants) | 6 | 0 | 6
Nanogram per milliliter
  GSK2391220 | 7.5219 (14.4) |  | 31.5278 (30.4)
  GSK2487818 | 6.0391 (19.1) |  | 25.4542 (33.0)
  GSK2506102 | 1.8233 (16.6) |  | 6.8139 (25.7)
  GSK2506104 | 7.3607 (13.5) |  | 30.4258 (27.6)
  GSK2531398 | 3.5279 (12.7) |  | 13.5590 (25.8)
  GSK2531401 | 6.4247 (23.6) |  | 21.9493 (36.8)

26. Secondary Outcome: Tmax of GSK1278863 Metabolites in Plasma Following Administration of IV and Both Oral Doses
Description: as for outcome 24
Time Frame: as for outcome 1
Population: as for outcome 23
Measure: Median (Full Range); unit: Hour
Arm/Group | GSK1278863 6 mg Oral Tablet | [14C]-GSK1278863 50 µg IV Infusion | [14C]-GSK1278863 25 mg Oral Solution
Number analyzed (Participants) | 6 | 0 | 6
Hour
  GSK2391220 | 3.5000 [2.983 to 6.000] |  | 2.0000 [1.500 to 4.000]
  GSK2487818 | 3.5000 [1.983 to 6.000] |  | 2.0000 [1.500 to 4.000]
  GSK2506102 | 3.5000 [2.983 to 6.000] |  | 2.0000 [2.000 to 4.000]
  GSK2506104 | 4.0000 [2.983 to 6.000] |  | 2.0000 [2.000 to 4.000]
  GSK2531398 | 3.5000 [2.983 to 6.000] |  | 2.0000 [2.000 to 4.000]
  GSK2531401 | 4.0000 [3.000 to 6.000] |  | 2.0000 [2.000 to 4.000]

27. Secondary Outcome: T1/2 of GSK1278863 Metabolites in Plasma Following Administration of IV and Both Oral Doses
Description: Plasma samples were collected from participants at indicated time points, for metabolite profiling. GSK2391220, GSK2506104, GSK2487818, GSK2506102, GSK2531398 and GSK2531401 were metabolites of GSK1278863. Pharmacokinetic analysis was conducted using standard non-compartmental methods. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles). Data were not collected for GSK1278863 metabolites following IV dose as analysis of pharmacokinetic parameters of only parent compound following IV dose was of interest to calculate the bioavailability and not the metabolites.
Time Frame: as for outcome 1
Population: as for outcome 23
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour
Arm/Group | GSK1278863 6 mg Oral Tablet | [14C]-GSK1278863 50 µg IV Infusion | [14C]-GSK1278863 25 mg Oral Solution
Number analyzed (Participants) | 6 | 0 | 6
Hour
  GSK2391220; n=6,0, 5: number analyzed (Participants) | 6 | 0 | 5
  GSK2391220; n=6,0, 5 | 1.9805 (7.9) |  | 3.1506 (26.1)
  GSK2487818; n=6,0, 6 | 1.5744 (12.5) |  | 1.8644 (10.7)
  GSK2506102; n=6,0, 6 | 2.0037 (15.9) |  | 2.2738 (5.1)
  GSK2506104; n=6,0, 5: number analyzed (Participants) | 6 | 0 | 5
  GSK2506104; n=6,0, 5 | 2.0849 (8.0) |  | 3.3870 (10.9)
  GSK2531398; n=6,0, 6 | 1.7006 (14.7) |  | 1.9767 (3.8)
  GSK2531401; n=6,0, 6 | 2.3217 (12.0) |  | 2.9197 (9.9)

28. Secondary Outcome: Vss of GSK1278863 in Plasma Following IV Dose Administration
Description: Plasma samples were collected from participants at indicated time points, after administration of radiolabeled IV dose of GSK1278863 to investigate the pharmacokinetics of GSK1278863 in plasma. Pharmacokinetic analysis was conducted using standard non-compartmental methods.
Time Frame: as for outcome 11
Population: Pharmacokinetic Population. Only those participants with data available at specified time point were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter
Arm/Group | [14C]-GSK1278863 50 µg IV Infusion
Number analyzed (Participants) | 3
Liter | 14.3387 (23.0)

29. Secondary Outcome: Vss of GSK1278863 Metabolites in Plasma Following IV Dose Administration
Description: Plasma samples were planned to be collected from participants at indicated time points, after administration of radiolabeled IV dose of GSK1278863 for metabolite profiling. GSK2391220, GSK2506104, GSK2487818, GSK2506102, GSK2531398 and GSK2531401 were metabolites of GSK1278863. Pharmacokinetic analysis was conducted using standard non-compartmental methods. Data were not collected for GSK1278863 metabolites following IV dose as analysis of pharmacokinetic parameters of only parent compound following IV dose was of interest to calculate the bioavailability and not the metabolites.
Time Frame: as for outcome 11
Population: as for outcome 23
Arm/Group | [14C]-GSK1278863 50 µg IV Infusion
Number analyzed (Participants) | 0

30. Secondary Outcome: CL of GSK1278863 in Plasma Following IV Dose Administration
Description: as for outcome 28
Time Frame: as for outcome 11
Population: Pharmacokinetic Population. Only those participants with data available at specified time point were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter per hour
Arm/Group | [14C]-GSK1278863 50 µg IV Infusion
Number analyzed (Participants) | 3
Liter per hour | 18.8612 (27.4)

31. Secondary Outcome: CL of GSK1278863 Metabolites in Plasma Following IV Dose Administration
Description: as for outcome 29
Time Frame: as for outcome 11
Population: as for outcome 23
Arm/Group | [14C]-GSK1278863 50 µg IV Infusion
Number analyzed (Participants) | 0

32. Secondary Outcome: Absolute Bioavailability of GSK1278863 Following Oral Dosing
Description: Absolute bioavailability is the amount of drug from a formulation that reaches the systemic circulation relative to an IV dose, computed as ratio of AUC(oral)/Dose(oral) with AUC(IV)/Dose(IV). Plasma samples were collected from participants at indicated time points. Absolute bioavailability from the oral tablet and IV doses administered in treatment period 1 was analyzed using AUC(0-inf) and AUC(0-t) pharmacokinetic parameters.
Time Frame: as for outcome 11
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of dose normalized AUC
Arm/Group | GSK1278863 6 mg Oral Tablet
Number analyzed (Participants) | 6
Ratio of dose normalized AUC
  AUC (0-inf); n=3: number analyzed (Participants) | 3
  AUC (0-inf); n=3 | 0.6575 (11.8)
  AUC (0-t); n=6 | 0.6263 (10.7)

33. Secondary Outcome: Percent Radioactivity Recovered for Each Metabolite in Plasma Following a Single Oral Dose of [14C]-GSK1278863 at 25 mg
Description: Blood samples were collected in treatment period 2 to measure total radioactivity and to characterize the metabolite profiling of GSK1278863 following a single oral dose of [14C]-GSK1278863 at 25 mg. Potential metabolites were M3 (GSK2506104), M2 (GSK2391220) and M33 combined, M4 (GSK2487818), M6 (GSK2531398), M13 (GSK2531401), M5 (GSK2506102) and M14 combined. 2 pooled plasma samples were prepared. Aliquots of plasma samples collected between 0 to 8 hours post-dose from each participant were pooled in proportion to the time intervals. An equal amount of the individual pools from each participant was then pooled to create 1 plasma sample that was representative of the mean area under curve over the range of 0-8 hour. The second pool (10-12 hours pool) was obtained by mixing equal volume of the plasma samples at 10 and 12 hour across all participants. Percent radioactivity recovered for each metabolite in plasma following a single oral dose of [14C]-GSK1278863 at 25 mg is presented.
Time Frame: 0-8 hours, 10-12 hours in period 2
Population: Pharmacokinetic Population
Measure: Number; unit: Percent radioactivity
Arm/Group | [14C]-GSK1278863 25 mg Oral Solution
Number analyzed (Participants) | 6
Percent radioactivity
  M2 (GSK2391220) and M33 combined, 0-8 hours | 10.4
  M2 (GSK2391220) and M33 combined, 10-12 hours | 14.4
  M3 (GSK2506104), 0-8 hours | 7.6
  M3 (GSK2506104), 10-12 hours | 11.8
  M4 (GSK2487818), 0-8 hours | 5.7
  M4 (GSK2487818), 10-12 hours | NA — Data is not available since concentration of metabolite was not detected in the sample.
  M6 (GSK2531398), 0-8 hours | 3.6
  M6 (GSK2531398), 10-12 hours | NA — Data is not available as all concentration values were less than the lower limit of quantification.
  M13 (GSK2531401), 0-8 hours | 8.3
  M13 (GSK2531401), 10-12 hours | 16.1
  M5 (GSK2506102) and M14 combined, 0-8 hours | 4.5
  M5 (GSK2506102) and M14 combined, 10-12 hours | NA — Data is not available as all concentration values were less than the lower limit of quantification.

34. Secondary Outcome: Percent Radioactivity Recovered for Each Metabolite in Urine Following a Single Oral Dose of [14C]-GSK1278863 at 25 mg
Description: Urine samples were collected in treatment period 2 to measure total radioactivity and to characterize the metabolite profiling of GSK1278863 following a single oral dose of [14C]-GSK1278863 at 25 mg. Potential metabolites were M3 (GSK2506104), M2 (GSK2391220) and M33 combined, M4 (GSK2487818), M6 (GSK2531398), M13 (GSK2531401), M5 (GSK2506102) and M14 combined. One pooled urine sample was prepared by urine collected from 0 to 24 hours post dose from all participants. Percent radioactivity recovered for each metabolite in urine following a single oral dose of [14C]-GSK1278863 at 25 mg is presented.
Time Frame: 0-24 hours in period 2
Population: Pharmacokinetic Population
Measure: Number; unit: Percent radioactivity
Arm/Group | [14C]-GSK1278863 25 mg Oral Solution
Number analyzed (Participants) | 6
Percent radioactivity
  M2 (GSK2391220) and M33 combined | 15.8
  M3 (GSK2506104) | 16.0
  M4 (GSK2487818) | 7.9
  M6 (GSK2531398) | 5.8
  M13 (GSK2531401) | 16.5
  M5 (GSK2506102) and M14 combined | 10.4

35. Secondary Outcome: Percent Radioactivity Recovered for Each Metabolite in Feces Following a Single Oral Dose of [14C]-GSK1278863 at 25 mg
Description: Feces samples were collected in treatment period 2 to measure total radioactivity and to characterize the metabolite profiling of GSK1278863 following a single oral dose of [14C]-GSK1278863 at 25 mg. Potential metabolites were M3 (GSK2506104), M2 (GSK2391220), M4 (GSK2487818), M6 (GSK2531398), M13 (GSK2531401), M5 (GSK2506102) and M14 combined. One pooled feces sample was prepared by samples collected from 0 to 120 hours post dose from all participants. Percent radioactivity recovered for each metabolite in feces following a single oral dose of [14C]-GSK1278863 at 25 mg is presented.
Time Frame: 0-120 hours in period 2
Population: Pharmacokinetic Population
Measure: Number; unit: Percent radioactivity
Arm/Group | [14C]-GSK1278863 25 mg Oral Solution
Number analyzed (Participants) | 6
Percent radioactivity
  M2 (GSK2391220) | 19.8
  M3 (GSK2506104) | 14.1
  M4 (GSK2487818) | 17.0
  M6 (GSK2531398) | 6.2
  M13 (GSK2531401) | 4.9
  M5 (GSK2506102) and M14 combined | 7.7

36. Secondary Outcome: Percent Radioactivity Recovered for Each Metabolite in Duodenal Bile Following a Single Dose of [14C]-GSK1278863 50 µg IV Infusion
Description: The bile string was swallowed by participants prior to oral dose and was removed 3 hours after the oral dose (1 hour after the end of the IV infusion) in treatment period-1. Duodenal bile string extracts were pooled to create a single pool sample to measure total radioactivity and to characterize the metabolite profiling of GSK1278863 following a single dose of [14C]-GSK1278863 50 µg IV infusion. Potential metabolites were M3 (GSK2506104), M2 (GSK2391220), M4 (GSK2487818), M6 (GSK2531398), M13 (GSK2531401), M5 (GSK2506102). Mean percent radioactivity recovered for each metabolite in bile following a single dose of [14C]-GSK1278863 50 µg IV infusion is presented.
Time Frame: 3 hours post-oral dose in period 1
Population: Pharmacokinetic Population. Only those participants with data available at specified time point were analyzed.
Measure: Number; unit: Percent radioactivity
Arm/Group | [14C]-GSK1278863 50 µg IV Infusion
Number analyzed (Participants) | 3
Percent radioactivity
  M2 (GSK2391220) | 12.3
  M3 (GSK2506104) | 20.0
  M4 (GSK2487818) | 15.5
  M6 (GSK2531398) | 6.3
  M13 (GSK2531401) | 2.4
  M5 | 11.1

37. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious AEs (SAEs)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the study treatment. A SAE is defined as any untoward medical occurrence that, at any dose which results in death, is life- threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity, is a congenital anomaly/birth defect, associated with liver injury and impaired liver function or any other situations as per Medical or scientific judgment. Safety Population comprised of all participants who take at least 1 dose of study treatment. Participants were analyzed according to the treatment they actually received.
Time Frame: Up to 43 days
Population: Safety Population
Measure: Count of Participants; unit: Participants
Groups:
- GSK1278863 6 mg Oral Tablet+[14C]-GSK1278863 50 µg IV Infusion: Participants received a single 6 mg oral dose of GSK1278863 on Day 1 of treatment period 1, after an overnight fast of at least 8 hours. After approximately 1 hour, participants received 50 µg [14C]-GSK1278863 by IV infusion over 1 hour.
Arm/Group | GSK1278863 6 mg Oral Tablet+[14C]-GSK1278863 50 µg IV Infusion | [14C]-GSK1278863 25 mg Oral Solution
Number analyzed (Participants) | 6 | 6
Participants
  Any AE | 2 | 2
  Any SAE | 0 | 0

38. Secondary Outcome: Number of Participants With AEs at a Particular Severity
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the study treatment. Severity was categorized as mild, moderate and severe. The number of participants with AEs at any type of severity (mild, moderate and severe) has been presented.
Time Frame: Up to 43 days
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1278863 6 mg Oral Tablet+[14C]-GSK1278863 50 µg IV Infusion | [14C]-GSK1278863 25 mg Oral Solution
Number analyzed (Participants) | 6 | 6
Participants
  Mild | 2 | 2
  Moderate | 1 | 0
  Severe | 0 | 0

39. Secondary Outcome: Number of Participants With Worst Case Clinical Chemistry Results Relative to Normal Range
Description: Blood samples were collected from participants at indicated time points for the analysis of clinical chemistry parameters including Alanine Aminotransferase (ALT), Alkaline phosphatase (Alk Phos), Aspartate Aminotransferase (AST), Bilirubin, Calcium, Creatinine, Direct Bilirubin, Glucose, Potassium, Protein, Sodium and Urea. Participants were counted in the worst case category that their value changes to (low, normal or high), unless there was no change in their category. Participants whose lab value category was unchanged (example given [e.g.], High to High), or whose value became normal, are recorded in the "To Normal or No Change" category. Participants were counted twice if the participant had values that changed 'To Low' and 'To High', so the percentages may not add to 100%. High and low indicated that the participants had values flagged as high and low respectively for the particular parameter any time on-treatment.
Time Frame: Up to 43 days
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1278863 6 mg Oral Tablet+[14C]-GSK1278863 50 µg IV Infusion | [14C]-GSK1278863 25 mg Oral Solution
Number analyzed (Participants) | 6 | 6
Participants
  ALT; To Low | 0 | 0
  ALT;To Normal or No Change | 6 | 6
  ALT; To High | 0 | 0
  Alk Phos; To Low | 0 | 0
  Alk Phos; To Normal or No Change | 6 | 6
  Alk Phos; To High | 0 | 0
  AST; To Low | 0 | 0
  AST;To Normal or No Change | 6 | 6
  AST; To High | 0 | 0
  Bilirubin; To Low | 0 | 0
  Bilirubin; To Normal or No Change | 5 | 6
  Bilirubin; To High | 1 | 1
  Calcium; To Low | 0 | 0
  Calcium; To Normal or No Change | 6 | 6
  Calcium; To High | 0 | 0
  Creatinine; To Low | 0 | 0
  Creatinine; To Normal or No Change | 6 | 6
  Creatinine; To High | 0 | 0
  Direct Bilirubin; To Low | 0 | 0
  Direct Bilirubin; To Normal or No Change | 6 | 6
  Direct Bilirubin; To High | 0 | 0
  Glucose; To Low | 0 | 0
  Glucose; To Normal or No Change | 6 | 6
  Glucose; To High | 0 | 0
  Potassium; To Low | 0 | 0
  Potassium; To Normal or No Change | 6 | 6
  Potassium; To High | 0 | 0
  Protein; To Low | 0 | 0
  Protein; To Normal or No Change | 6 | 6
  Protein; To High | 0 | 0
  Sodium; To Low | 1 | 0
  Sodium; To Normal or No Change | 5 | 6
  Sodium; To High | 0 | 0
  Urea; To Low | 0 | 0
  Urea;To Normal or No Change | 6 | 6
  Urea; To High | 0 | 0

40. Secondary Outcome: Number of Participants With Worst Case Hematology Results Relative to Normal Range
Description: Blood samples were collected from participants at indicated time points for the analysis of hematology parameters including Basophils, Eosinophils, Erythrocyte Mean Corpuscular Hemoglobin (MCH), Erythrocyte Mean Corpuscular Volume (MCV), Erythrocytes, Hematocrit, Hemoglobin, Leukocytes, Lymphocytes, Monocytes, Neutrophils, Platelets, Reticulocytes, and Reticulocytes/Erythrocytes. Participants were counted in the worst case category that their value changes to (low, normal or high), unless there was no change in their category. Participants whose lab value category was unchanged (e.g., High to High), or whose value became normal, are recorded in the "To Normal or No Change" category. Participants were counted twice if the participant had values that changed 'To Low' and 'To High', so the percentages may not add to 100%. High and low indicated that the participants had values flagged as high and low respectively for the particular parameter any time on-treatment.
Time Frame: Up to 43 days
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1278863 6 mg Oral Tablet+[14C]-GSK1278863 50 µg IV Infusion | [14C]-GSK1278863 25 mg Oral Solution
Number analyzed (Participants) | 6 | 6
Participants
  Basophils; To Low | 0 | 0
  Basophils; To Normal or No Change | 6 | 6
  Basophils; To High | 0 | 0
  Eosinophils; To Low | 0 | 0
  Eosinophils; To Normal or No Change | 6 | 6
  Eosinophils; To High | 0 | 0
  MCH; To Low | 0 | 0
  MCH; To Normal or No Change | 6 | 6
  MCH; To High | 0 | 0
  MCV; To Low | 0 | 0
  MCV; To Normal or No Change | 6 | 6
  MCV; To High | 0 | 0
  Erythrocytes; To Low | 1 | 0
  Erythrocytes; To Normal or No Change | 5 | 6
  Erythrocytes; To High | 0 | 0
  Hematocrit; To Low | 1 | 1
  Hematocrit; To Normal or No Change | 5 | 5
  Hematocrit; To High | 0 | 0
  Hemoglobin; To Low | 1 | 0
  Hemoglobin; To Normal or No Change | 5 | 6
  Hemoglobin; To High | 0 | 0
  Leukocytes; To Low | 0 | 0
  Leukocytes; To Normal or No Change | 6 | 6
  Leukocytes; To High | 0 | 0
  Lymphocytes; To Low | 1 | 0
  Lymphocytes; To Normal or No Change | 5 | 6
  Lymphocytes; To High | 0 | 0
  Monocytes; To Low | 0 | 0
  Monocytes; To Normal or No Change | 6 | 6
  Monocytes; To High | 0 | 0
  Neutrophils; To Low | 0 | 0
  Neutrophils; To Normal or No Change | 6 | 6
  Neutrophils; To High | 0 | 0
  Platelets; To Low | 0 | 0
  Platelets; To Normal or No Change | 6 | 6
  Platelets; To High | 0 | 0
  Reticulocytes; To Low | 0 | 0
  Reticulocytes; To Normal or No Change | 6 | 6
  Reticulocytes; To High | 0 | 1
  Reticulocytes/Erythrocytes; To Low | 0 | 0
  Reticulocytes/Erythrocytes; To Normal or No Change | 6 | 5
  Reticulocytes/Erythrocytes; To High | 0 | 2

41. Secondary Outcome: Number of Participants With Abnormal Urinalysis Findings
Description: Urine samples were collected at indicated time points for the analysis of urinalysis parameters including specific gravity and PH of urine, presence of glucose, protein, blood, ketones, bilirubin, urobilinogen, nitrite, leukocyte esterase in urine.
Time Frame: Up to 43 days
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1278863 6 mg Oral Tablet+[14C]-GSK1278863 50 µg IV Infusion | [14C]-GSK1278863 25 mg Oral Solution
Number analyzed (Participants) | 6 | 6
Participants | 0 | 0

42. Secondary Outcome: Number of Participants With Abnormal Electrocardiogram (ECG) Findings
Description: Full 12-lead ECGs were recorded with the participant in a supine position. The number of participants with abnormal ECG findings at indicated time points were presented. Data has been presented for participants with respect to the actual treatment received in respective treatment periods.
Time Frame: Pre-dose (on Day 1) and Day 8 in treatment period 2; 144 hours (Day 7) in treatment period 1
Population: Safety Population. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1278863 6 mg Oral Tablet+[14C]-GSK1278863 50 µg IV Infusion | [14C]-GSK1278863 25 mg Oral Solution
Number analyzed (Participants) | 6 | 6
Participants
  Pre-dose (Day 1); n=0,6: number analyzed (Participants) | 0 | 6
  Pre-dose (Day 1); n=0,6 |  | 0
  144 hours (Day 7); n= 6, 0: number analyzed (Participants) | 6 | 0
  144 hours (Day 7); n= 6, 0 | 0 |
  Day 8; n=0, 6: number analyzed (Participants) | 0 | 6
  Day 8; n=0, 6 |  | 0

43. Secondary Outcome: Change From Baseline in Blood Pressure
Description: Vital sign including systolic and diastolic blood pressure were measured in a semi-supine position after 5 minutes rest. Baseline is defined as the mean of the 3 pre-dose measurements (Average [Avg] Pre-dose) taken on Day 1 in each treatment period. Change from Baseline was defined as any visit value minus the Baseline value. Data has been presented for participants with respect to the actual treatment received in respective treatment periods.
Time Frame: Baseline (average of Pre-dose on Day 1 in treatment period 1 and 2); 3 hours, 144 hours (Day 7) in treatment period 1; 3 hours, 144 hours (Day 7) and Day 8 in treatment period 2
Population: as for outcome 42
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | GSK1278863 6 mg Oral Tablet+[14C]-GSK1278863 50 µg IV Infusion | [14C]-GSK1278863 25 mg Oral Solution
Number analyzed (Participants) | 6 | 6
Millimeters of mercury
  SBP; Avg 3 hours; n=6, 6 | -0.17 (5.722) | -1.22 (3.468)
  SBP; Avg 144 hours (Day 7); n=6, 6 | 5.06 (10.521) | -2.00 (9.541)
  SBP; Avg Day 8; n=0,6: number analyzed (Participants) | 0 | 6
  SBP; Avg Day 8; n=0,6 |  | 4.22 (4.075)
  DBP; Avg 3 hours; n=6, 6 | 1.22 (5.484) | 0.89 (4.834)
  DBP; Avg 144 hours (Day 7); n=6, 6 | 3.61 (9.365) | -1.00 (9.814)
  DBP; Avg Day 8; n=0,6: number analyzed (Participants) | 0 | 6
  DBP; Avg Day 8; n=0,6 |  | 3.39 (5.170)

44. Secondary Outcome: Change From Baseline in Heart Rate
Description: Heart rate was measured in a semi-supine position after 5 minutes rest. Baseline is defined as the mean of the 3 pre-dose measurements (Avg Pre-dose) taken on Day 1 in each treatment period. Change from Baseline was defined as any visit value minus the Baseline value. Data has been presented for participants with respect to the actual treatment received in respective treatment periods.
Time Frame: as for outcome 43
Population: as for outcome 42
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | GSK1278863 6 mg Oral Tablet+[14C]-GSK1278863 50 µg IV Infusion | [14C]-GSK1278863 25 mg Oral Solution
Number analyzed (Participants) | 6 | 6
Beats per minute
  Avg 3 hours; n=6, 6 | 0.22 (3.526) | 1.67 (3.425)
  Avg 144 hours (Day 7); n=6, 6 | 1.28 (6.571) | 3.78 (5.500)
  Avg Day 8; n=0,6: number analyzed (Participants) | 0 | 6
  Avg Day 8; n=0,6 |  | 4.72 (5.535)

45. Secondary Outcome: Change From Baseline in Respiratory Rate
Description: Respiratory rate was measured in a semi-supine position after 5 minutes rest. Baseline is defined as the pre-dose on Day 1 in each treatment period. Change from Baseline was defined as any visit value minus the Baseline value. Data has been presented for participants with respect to the actual treatment received in respective treatment periods.
Time Frame: Baseline (Pre-dose on Day 1 in treatment period 1 and 2); 3 hours, 144 hours (Day 7) in treatment period 1; 3 hours, 144 hours (Day 7) and Day 8 in treatment period 2
Population: as for outcome 42
Measure: Mean (Standard Deviation); unit: Breaths per minute
Arm/Group | GSK1278863 6 mg Oral Tablet+[14C]-GSK1278863 50 µg IV Infusion | [14C]-GSK1278863 25 mg Oral Solution
Number analyzed (Participants) | 6 | 6
Breaths per minute
  3 hours; n=6, 6 | -0.67 (2.422) | -0.33 (4.082)
  144 hours (Day 7); n=6, 6 | -1.33 (2.066) | -0.33 (1.506)
  Day 8; n=0,6: number analyzed (Participants) | 0 | 6
  Day 8; n=0,6 |  | 0.00 (2.530)

46. Secondary Outcome: Change From Baseline in Body Temperature
Description: Body temperature measurement was performed in participants at indicated time points. Baseline is defined as the pre-dose on Day 1 in each treatment period. Change from Baseline was defined as any visit value minus the Baseline value. Data has been presented for participants with respect to the actual treatment received in respective treatment periods.
Time Frame: as for outcome 45
Population: as for outcome 42
Measure: Mean (Standard Deviation); unit: Celsius
Arm/Group | GSK1278863 6 mg Oral Tablet+[14C]-GSK1278863 50 µg IV Infusion | [14C]-GSK1278863 25 mg Oral Solution
Number analyzed (Participants) | 6 | 6
Celsius
  3 hours; n=6, 6 | 0.08 (0.183) | 0.25 (0.455)
  144 hours (Day 7); n=6, 6 | 0.07 (0.446) | 0.12 (0.588)
  Day 8; n=0,6: number analyzed (Participants) | 0 | 6
  Day 8; n=0,6 |  | 0.30 (0.693)

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious adverse events (Non-SAEs) were collected from the start of the study treatment up to 43 days.
Description: SAEs and Non-SAEs were reported by treatment for the Safety Population which comprised of all participants who had taken at least 1 dose of study treatment
Arm/Group | GSK1278863 6 mg Oral Tablet+[14C]-GSK1278863 50 µg IV Infusion | [14C]-GSK1278863 25 mg Oral Solution
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 2/6 | 2/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK1278863 6 mg Oral Tablet+[14C]-GSK1278863 50 µg IV Infusion (N=6) | [14C]-GSK1278863 25 mg Oral Solution (N=6)
Headache (Nervous system disorders) | 1 (1) | 1 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-09-01): https://cdn.clinicaltrials.gov/large-docs/22/NCT03239522/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-30): https://cdn.clinicaltrials.gov/large-docs/22/NCT03239522/SAP_001.pdf